CLINICAL TRIAL: NCT03216564
Title: Intervention Using Vitamin D for Elevated Urinary ALbumin in Diabetes (IDEAL-2)
Brief Title: An Intervention to Examine the Effect of Vitamin D on Urine Protein Levels in Type 2 Diabetes
Acronym: IDEAL-2
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hamad Medical Corporation (Industry)
Collaborators: Weill Cornell Medical College in Qatar (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 16235/16; 1400039 (Other: Weill Cornell Medicine - Qatar)
Record Dates: First submitted 2017-06-19; First posted 2017-07-13 (Actual); Last update posted 2018-09-06 (Actual); Status verified 2018-07

CONDITIONS: Diabetic Nephropathies
MeSH Terms: conditions — Diabetic Nephropathies | interventions — Calcitriol

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Group (Experimental): Participants are treated with angiotensin converting enzyme inhibitor/angiotensin receptor blocker (ACEI/ARB) AND active vitamin D (Calcitriol) 0.25 micrograms orally per day for 26 weeks.
  Interventions: Drug: Calcitriol
- Usual Care (No Intervention): Participants are treated with ACEI/ARB alone for 26 weeks.

INTERVENTIONS:
Drug: Calcitriol — Active vitamin D (Calcitriol) 0.25 micrograms
  Other Names: Active Vitamin D
  Arms: Intervention Group

SUMMARY:
Diabetic kidney disease (nephropathy) develops in nearly 40% of patients with type 2 diabetes mellitus. Diabetic nephropathy is caused by damage to the small blood vessels in the kidneys due to uncontrolled blood sugar levels, which mean that the kidneys become less effective at filtering urine. This is associated with albuminuria (protein in the urine). Treatment with some drugs reduces the loss of albumin through the urine and delays disease progression. There is increasing evidence that vitamin D could also be important in management of diabetic kidney disease. The aim of this study is to investigate the efficacy and safety of a combined regimen of calcitriol (active vitamin D) and established drugs for diabetic kidney disease.

DETAILED DESCRIPTION:
The investigators propose to test the efficacy and safety of a combined regimen of calcitriol and angiotensin converting enzyme inhibitor (ACEI) or angiotensin receptor blocker (ARB) in type 2 diabetes subjects with albuminuria. In the proposed study, the bioactive form of vitamin D (calcitriol) is being used for its ability to synergize with ACEI or ARB and prevent renal disease progression. The study expands on preliminary studies demonstrating a reduction in proteinuria with vitamin D analogue treatment, in subjects with both diabetic as well as non-diabetic kidney disease.

ELIGIBILITY:
Inclusion Criteria:

1. Age greater than or equal to 18 years and less than 80 years
2. Diagnosis of T2DM requiring treatment with at least one oral hypoglycaemic medication or insulin 2.1. Subjects will be considered to have established T2DM if the diagnosis of diabetes has been made and the subjects were treated with insulin or an oral hypoglycaemic agent for at least 6 months after diagnosis 2.2. Subjects will be considered to have newly established T2DM if the diagnosis of diabetes was diagnosed with a fasting plasma glucose ≥ 7 mmol/L (126 mg/dL) or haemoglobin A1c is >6.5% in the past 6 months
3. Documented albuminuria defined as a presence of albuminuria on two occasions in the last six months:

   3.1. Albumin ≥ 30 mg/24 hour in a 24 hour urine collection, or 3.2. Albumin ≥ 20 μg/min in a short-time urine collection, or 3.3. Albumin ≥ 30 mg/L in a spot urine sample, or 3.4. A spot-urine albumin-creatinine ration (ACR) ≥ 30 mg/g creatinine (≥ 2.5 mg/mmol creatinine in men, ≥ 3.5 mg/mmol creatinine in women)
4. Estimated glomerular filtration rate (eGFR) using the 4-variable Modification of Diet in Renal Disease (MDRD) equation of ≥ 25 mL/min/1.73 m2

Exclusion Criteria:

1. If female, positive pregnancy test or planning pregnancy in the subsequent 12 months
2. Pregnant
3. Breastfeeding
4. Corrected serum calcium ≥ 2.62 mmol/L
5. Serum Potassium > 5.2 mmol/L if not on ACEI or ARB; Serum Potassium > 6.0 mmol/L if on ACEI or ARB
6. 25-hydroxyvitamin D (25-OH Vit D) > 80 ng/mL
7. PTH > 200 pg/mL
8. Poorly controlled hypertension defined as systolic blood pressure ≥ 180 mm Hg or diastolic blood pressure ≥ 110 mm Hg
9. Systolic blood pressure (SBP) ≤ 110 mm Hg
10. History of kidney stones
11. History of severe chronic disease (e.g. chronic liver disease)
12. Active malignancy
13. Recent diagnosis of acute renal failure within 3 months of screening visit
14. Likelihood of renal replacement therapy within 1 year

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 320 (Estimated)
Dates: Start 2017-05-10 (Actual); Primary Completion 2019-05-10 (Estimated); Study Completion 2019-05-10 (Estimated)

PRIMARY OUTCOMES:
Urinary albumin creatinine ratio (ACR) measured biochemically | 26 weeks
  Urine albumin and creatinine will be measured biochemically and their ratio calculated

SECONDARY OUTCOMES:
24-hour urine albumin (24h UA) excretion | 26 weeks
  24-hour urine albumin (24h UA) excretion measured biochemically
Estimated glomerular filtration rate (eGFR) | 26 weeks
  Calculated using the Modification of Diet in Renal Disease (MDRD) equation
Blood pressure | 26 weeks
  Blood pressure measured using a digital sphygmomanometer

OTHER OUTCOMES:
Patient Reported Outcome: Quality of life | 26 weeks
  Measured using the EQ5D questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Muhammad Asim, MB BS, Principal Investigator — Hamad Medical Corporation
Locations (1):
- Hamad Medical Corporation, Doha, Qatar

IPD SHARING:
Plan to Share IPD: Undecided
For data, please contact investigators

REFERENCES:
- [Derived] Taheri S, Asim M, Al Malki H, Fituri O, Suthanthiran M, August P; IDEAL-2 Study Team. Intervention using vitamin D for elevated urinary albumin in type 2 diabetes mellitus (IDEAL-2 Study): study protocol for a randomised controlled trial. Trials. 2018 Apr 17;19(1):230. doi: 10.1186/s13063-018-2616-5. PMID 29665833